CLINICAL TRIAL: NCT07136116
Title: A Prospective, Real-World Study Evaluating the Impact of RISankizumab on BurdEn of Disease in Ulcerative Colitis in JaPan (RISE UP)
Brief Title: Study to Assess Change in Disease Activity of Risankizumab Treatment in Japanese Participants With Moderate to Severe Ulcerative Colitis
Acronym: RISE UP
Status: Recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P25-797
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis; Risankizumab; SKYRIZI
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Risankizumab: Participants will receive risankizumab as prescribed by their physician according to local label.

SUMMARY:
Ulcerative colitis (UC) is a type of inflammatory bowel disease that causes inflammation and bleeding from the lining of the rectum and colon (large intestine). This study will assess the change in disease activity of risankizumab treatment in adult participants with moderate to severe UC in real-world clinical practice.

Risankizumab is an approved drug for treating participants with ulcerative colitis. Approximately 200 participants who are prescribed risankizumab by their physician in accordance with local label will be enrolled in approximately 30 sites across Japan.

Participants will receive risankizumab as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for up to 156 weeks.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with a diagnosis of moderate to severe Ulcerative Colitis (UC) commenced on Risankizumab (RZB) treatment prescribed as part of their routine clinical care at their clinical's discretion according to Japan approved label and treatment prescription recommendations/guidelines.
* The decision to prescribe RZB is made prior to and independently of study participation.
* Participants able to provide voluntary informed consent before any study-related activities or procedures (obtained/documented as per regulations). If the patient is under 18 years old, a patient's parent or legal guardian must be willing to give written informed consent.
* Participants who can understand and communicate with the investigator and comply with the requirements of the study, including collection of PRO data using a smart device (i.e., mobile phone) and continued PRO data collection after cessation of RZB.
* Participants without previous exposure to RZB.
* Participants who are not currently participating in interventional research (not including non-interventional studies, PMOS, or registry participation).

Exclusion Criteria:

See Inclusion Criteria

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include adult participants with moderate to severe UC who are being treated with RZB according to the relevant approved license and who are eligible according to the study eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
To assess the achievement of clinical remission per Partial Adapted Mayo Score of Risankizumab treatment in participants with moderate to severe Ulcerative Colitis (UC) | At Week 52
  Defined as stool frequency subscore [SFS] ≤1 and rectal bleeding subscore [RBS]=0

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (25):
- Japan (25):
  - Aichi Medical University Hospital /ID# 278155, Nagakute, Aichi-ken
  - Nagoya University Hospital /ID# 278159, Nagoya, Aichi-ken
  - Hirosaki University Hospital /ID# 278153, Hirosaki, Aomori
  - Chiba University Hospital /ID# 277669, Chiba, Chiba
  - Tsujinaka Hospital - Kashiwanoha /ID# 277672, Kashiwa-shi, Chiba
  - Toho University Sakura Medical Center /ID# 277536, Sakura, Chiba
  - Kyushu University Hospital /ID# 278077, Fukuoka, Fukuoka
  - Sapporo Medical University Hospital /ID# 277535, Sapporo, Hokkaido
  - Hokkaido University Hospital /ID# 277668, Sapporo, Hokkaido
  - Sapporo Higashi Tokushukai Hospital /ID# 278123, Sapporo, Hokkaido
  - Kobe University Hospital /ID# 278292, Kobe, Hyōgo
  - Hyogo Medical University Hospital /ID# 277676, Nishinomiya-shi, Hyōgo
  - University Hospital Kyoto Prefectural University of Medicine /ID# 277541, Kyoto, Kyoto
  - Kansai Medical University Hospital /ID# 278619, Hirakata-shi, Osaka
  - Saga University Hospital /ID# 278160, Saga, Saga-ken
  - Saitama Medical Center /ID# 278076, Kawagoe, Saitama
  - Shiga University of Medical Science Hospital /ID# 277540, Ōtsu, Shiga
  - Hamamatsu University Hospital /ID# 277539, Hamamatsu, Shizuoka
  - NHO Shizuoka Medical Center /ID# 278075, Sunto-gun, Shizuoka
  - Dokkyo Medical University Hospital /ID# 278152, Mibu, Tochigi
  - Institute of Science Tokyo Hospital /ID# 277538, Bunkyo-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital /ID# 278154, Minato-ku, Tokyo
  - Kyorin University Hospital /ID# 277534, Mitaka-shi, Tokyo
  - Fukuoka University Hospital /ID# 277677, Fukuoka
  - Sapporo Kosei General Hospital /ID# 278048, Sapporo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P25-797